CLINICAL TRIAL: NCT06398990
Title: The Effect of Telerehabilitation-Based Cognitive Exercise Therapy Approach and Yoga on Pain, Physical Function and Quality of Life in Adolescents With Dysmenorrhoea
Brief Title: The Effect of Cognitive Exercise Therapy Approach and Yoga in Adolescents With Dysmenorrhoea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Dilek Cagri, Principal Investigator, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1/35
Record Dates: First submitted 2024-04-03; First posted 2024-05-03 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-01

CONDITIONS: Dysmenorrhea; Primary Dysmenorrhea
Keywords: dysmenorrhea; mind-body exercises; cognitive exercise therapy approach; yoga
MeSH Terms: conditions — Dysmenorrhea | interventions — Yoga

STUDY DESIGN:
Masking Description: Because the study involved mind-body exercise practices such as cognitive exercise therapy approach and yoga, and because participants directly experienced the type of exercise, it was impossible to conceal which group they were in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Exercise Therapy Approach (Experimental): Cognitive exercise therapy sessions will consist of exercises including various movements in one session and the exercises will be worked with respiratory control, accompanied by a physiotherapist.
  Interventions: Other: Cognitive Exercise Therapy Approach
- Yoga Programme (Experimental): Yoga sessions will consist of exercises including various movements in one session and the exercises will be practised with respiratory control, accompanied by a physiotherapist.
  Interventions: Other: Yoga
- Routine Medical Treatment (Other): Individuals in this group will receive medical treatment recommended by the relevant physician.
  Interventions: Other: Routine Medical Treatment

INTERVENTIONS:
Other: Cognitive Exercise Therapy Approach — It will continue twice a week for 12 weeks. After the initial evaluation of the cases, one-on-one, face-to-face training will be provided with the patient in the first week (2 sessions) in order to ensure their compliance with the treatment and to fully understand the treatment method. Then, treatments will be carried out synchronously with the patients twice a week via the online platform (Zoom).
  Arms: Cognitive Exercise Therapy Approach
Other: Yoga — It will continue twice a week for 12 weeks. After the initial evaluation of the cases, one-on-one, face-to-face training will be provided with the patient in the first week (2 sessions) in order to ensure their compliance with the treatment and to fully understand the treatment method. Then, treatments will be carried out synchronously with the patients twice a week via the online platform (Zoom).
  Arms: Yoga Programme
Other: Routine Medical Treatment — Assessments of individuals in this group will be made face-to-face in the relevant clinic.
  Arms: Routine Medical Treatment

SUMMARY:
Dysmenorrhoea is a condition that negatively affects the quality of life in women of many age groups. In girls with dysmenorrhoea in adolescence, there is an effect on school performance, self-confidence-depression problems and a decrease in quality of life due to pain. In order to eliminate these negative effects, they should receive a good treatment. Medical treatment usually tries to minimise and balance this situation. Considering the fact that families do not want to use drugs such as oral contraceptives in their children at this age and the risks of oral contraceptives, parents are in different searches. Considering that the approach to pain should always be from a holistic perspective, yoga and cognitive exercise therapy approaches are both biopsychosocial treatment methods within the scope of mind-body integrity. Yoga and cognitive exercise therapy approach is thought to reduce symptoms, improve physical functions and quality of life in adolescent girls. With these positive effects, school absenteeism decreases, depression and self-confidence improve. Health costs will also be reduced to some extent.

DETAILED DESCRIPTION:
This study was designed as a prospective, randomised, controlled, parallel group study.

G-Power Statistical and Qualitative Data Analysis Software version 3.1.9.2 will be used to estimate the sample size required for the study. Considering that the study consists of a total of three parallel groups (cognitive exercise therapy approach, yoga, control) with measurements taken at three different time points, and given an effect size of Cohen's f = 0.25 and a significance level (α) of 0.05, and power (1-β error level) of 0.80, the total sample size is planned to be 36 cases, with a minimum of 12 cases per group. Considering a potential follow-up loss rate of 20%, it is estimated that at least 42 participants should be included in the study.

In similar studies in the literature, the effect size observed in menstrual pain levels is very large. Considering that the effect size may be more moderate in real life and in order to increase the publishability of the research findings, the effect size was set to Cohen's f = 0.25 and the sample size calculation was performed.

The 1st intervention group will receive cognitive exercise therapy approach, the 2nd intervention group will receive yoga, and the 3rd control group will consist of people receiving routine medical treatment. In order to fully reveal the effectiveness of the applications, reduce bias, and ensure homogeneity between the training and control groups, the distribution of groups will be determined randomly using a computer program.

Yoga and cognitive exercise therapy approach will be applied by a physiotherapist who has training in both fields. Treatments will continue twice a week for 12 weeks. After the initial assessment of the cases, one-to-one, face-to-face trainings will be carried out in the first week (2 sessions) in order to ensure their compliance with the treatment and to fully understand the treatment method. Afterwards, treatments will be carried out synchronously with the patients 2 times a week via the online platform.

Evaluations will be carried out 3 times as pre-treatment, 6th week and 12th week. All evaluations will be made face-to-face in the relevant clinic.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 10 and 19,
* Having had a menstrual cycle for at least 6-12 months (ACOG, 2018),
* Having menstrual pain intensity of ≥4 cm according to the Visual Analog Scale (VAS, 0-10 cm) (Kannan, P. 2015; Yonglitthipagon, P. 2017),
* To have been diagnosed with primary dysmenorrhea according to the clinical characteristics and diagnostic approach defined in international dysmenorrhea guidelines (ACOG 2018; JOGC 2017),
* Nulliparous (having never given birth),
* Able to read and write in Turkish,
* Willing to participate in the study and having provided informed consent.

Exclusion Criteria:

* History or clinical findings suggestive of secondary dysmenorrhea,
* Presence of serious comorbidities, including neurological, cardiovascular, musculoskeletal, psychiatric, gastrointestinal, or autoimmune disorders,
* History of surgery involving the abdominal, pelvic, or spinal regions within the past 12 months,
* Current pregnancy or suspected pregnancy,
* Use of intrauterine devices (IUDs),
* Current or recent participation in cognitive exercise therapy and/or yoga interventions,
* Concurrent participation in another clinical study.

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (VAS) | Pain intensity will be assessed 2 days before, 1 day before, on the 1st, 2nd and 3rd day of menstruation.
  In the 10 cm VAS, which is the most widely used, reliable and valid scale in the evaluation of pain intensity all over the world, the left end of the line will be formed as "0 = no pain" and the other end as "10 = unbearable pain". The subjects will be given paper in the form of a pain diary to mark during their menstrual periods and will be asked to mark the point appropriate to the intensity of pain 2 days before, 1 day before, on the 1st, 2nd and 3rd day of menstruation.
Physical function (Flexibility) | It will be done 3 times: before the treatment, at the 6th week and at the 12th week.
  Sit-Reach Test: The flexibility of the subjects participating in the study will be evaluated with a standard sit-and-reach box (Sit and Reach Trunk Flexibility Assessment Testing Box, Baseline, NY, USA).
Physical function (Peripheral muscle strength) | It will be done 3 times: before the treatment, at the 6th week and at the 12th week.
  Peripheral Muscle Strength: To evaluate the peripheral muscle strength of the subjects, hip flexors, hip extensors and hip abductors will be evaluated with a hand-held dynamometer in both legs.
Physical function (Respiratory Function) | It will be done 3 times: before the treatment, at the 6th week and at the 12th week.
  Respiratory Function: Pulmonary function tests are easy and reliable for evaluating and monitoring the effects of treatment on respiratory function. Spirometry is commonly used to assess respiratory function for this purpose. Measurements will be performed in accordance with American Thoracic Society (ATS)/European Respiratory Society (ERS) standards. FVC, FEV1, FEV1/FVC, and peak expiratory flow (PEF) parameters will be measured and recorded.
Physical function (Heart Rate Variability) | It will be done 3 times: before the treatment, at the 6th week and at the 12th week.
  Heart Rate Variability: Heart rate variability (HRV) defines the autonomic modulation of heart rate. It reflects parasympathetic activity and sympathetic/parasympathetic nervous system balance. Neuroimaging studies have shown that nociceptive stimulation is closely related to autonomic nervous system activity. Pain can cause a decrease in parasympathetic activity, an increase in sympathetic activity, and sympathovagal imbalance. Autonomic nervous system imbalance caused by sympathetic overactivity may be another cause of primary dysmenorrhea. In response to changes in the external environment, the ANS maintains homeostasis of the internal environment of the human body through the interaction between the sympathetic and parasympathetic nerves. A lack of coordination between the two systems can cause various symptoms. For these reasons, heart rate variability will be measured and recorded in adolescent girls with primary dysmenorrhea using the Polar H10 device.
Adolescent quality of life | It will be done 3 times: before the treatment, at the 6th week and at the 12th week.
  Pediatric Quality of Life Inventory TM (PedsQL)(Adolescent Form): The PedsQL is a quality of life scale that is suitable for use in both healthy and diseased children and adolescents. The PedsQL consists of child and parent forms aged 2-18 years. Since the adolescent group will be included in this study, the 13-18 years old Adolescent Form will be used. Scoring is done in 3 areas. Firstly, the total scale score (TSS), secondly, the total physical health score (PHSS), and thirdly, the total psychosocial health score (TPHSS), which consists of the calculation of item scores evaluating emotional, social and school functionality, are calculated. The items are scored between 0-100. If the answer to the question is marked as never, 100 points are scored; if it is marked as rarely, 75 points are scored; if it is marked as sometimes, 50 points are scored; if it is marked as frequently, 25 points are scored; if it is marked as almost always, 0 points are scored.

SECONDARY OUTCOMES:
Education absenteeism | It will be done twice: before the treatment and at the 12th week after the treatment.
  Adolescents with dysmenorrhea are typically of school age and may miss several days of school due to dysmenorrhea experienced during their menstrual periods. Therefore, the school absences of participants in the study will be monitored throughout the process. School absence rates before and after treatment will be compared.
Depression, anxiety, stress level | It will be done 3 times: before the treatment and 12 weeks after the treatment.
  Depression-Anxiety-Stress Scale Short Form (DASS-21): Both the original 42-item version of the DASS and the shorter 21-item version have been shown to be reliable and valid scales for measuring depression, anxiety and stress levels, through studies conducted with clinical groups, society and different cultural and ethnic groups. 7 items of DASS-21 include questions about depression, 7 items about anxiety, and 7 items about stress. Each subscale (depression, anxiety, stress) has a minimum of 0 and a maximum of 21 points. A low score indicates a good psychological state.
Dysmenorrhea Impact | It will be done 3 times: before the treatment and 12 weeks after the treatment.
  Revised Dysmenorrhea Impact Scale-Short Form (DIS-R): This 13-item scale, which includes cognitive/emotional (8 items) and physiological (5 items) subscales, has been shown to be a valid and reliable measurement tool. The minimum score on the scale is 0 and the maximum score is 65. As the scores increase, the functional and emotional impact level of individuals with dysmenorrhea also increases.
Physical activity | It will be done 3 times: before the treatment and 12 weeks after the treatment.
  Physical Activity Questionnaire for Adolescents (PAQ-A): Designed to provide a general estimate of physical activity levels among healthy adolescents, assessing sports participation and activities during and after school, self-administered and based on the last week. Later, a modified form for adolescents was published. The Turkish validity and reliability study of the scale was conducted. 8 questions in the scale are scored between 1 and 5, and the 9th question questions the presence of a condition that prevents physical activity during the last week. A score of '1' corresponds to low-intensity physical activity and a score of '5' corresponds to high-intensity physical activity, but the last question is not included in the scoring. The total score is obtained by calculating the average score of all questions.
Patient satisfaction | It will be done twice: before the treatment and at the 12th week after the treatment.
  The question of whether a patient is improving is fundamental in clinical practice, and the information obtained is important in making decisions regarding prognosis and treatment. Global Rating of Change (GROC) scales are widely used in clinical research, especially in the field of the musculoskeletal system. These scales are a rapid, effective method designed to measure a patient's improvement or worsening over time, usually either to determine the effect of an intervention or to chart the clinical course of a condition.
  In our study, to measure treatment satisfaction, "-2" means "I am very bad compared to before treatment", "-1" means "I am worse than before treatment", "0" means there is no change compared to before treatment, "1" means I am better than before treatment, "2" means I am very better than before treatment. The Global Rating of Change (GROC) scale will be used in the five-point Likert system.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Çağrı Arslan, Lecturer, Principal Investigator — Acıbadem Mehmet Ali Aydınlar University
Locations (1):
- Acibadem Mehmet Ali Aydinlar University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
At the end of the study, the general data results of the participants will be given statistically. Individual data sets will not be shared.

REFERENCES:
- [Background] Gutman G, Nunez AT, Fisher M. Dysmenorrhea in adolescents. Curr Probl Pediatr Adolesc Health Care. 2022 May;52(5):101186. doi: 10.1016/j.cppeds.2022.101186. Epub 2022 May 4. PMID 35523674
- [Background] Unnisa H, Annam P, Gubba NC, Begum A, Thatikonda K. Assessment of quality of life and effect of non-pharmacological management in dysmenorrhea. Ann Med Surg (Lond). 2022 Aug 30;81:104407. doi: 10.1016/j.amsu.2022.104407. eCollection 2022 Sep. PMID 36147090
- [Background] De Sanctis V, Soliman A, Bernasconi S, Bianchin L, Bona G, Bozzola M, Buzi F, De Sanctis C, Tonini G, Rigon F, Perissinotto E. Primary Dysmenorrhea in Adolescents: Prevalence, Impact and Recent Knowledge. Pediatr Endocrinol Rev. 2015 Dec;13(2):512-20. PMID 26841639
- [Background] Ferries-Rowe E, Corey E, Archer JS. Primary Dysmenorrhea: Diagnosis and Therapy. Obstet Gynecol. 2020 Nov;136(5):1047-1058. doi: 10.1097/AOG.0000000000004096. PMID 33030880
- [Background] Yonglitthipagon P, Muansiangsai S, Wongkhumngern W, Donpunha W, Chanavirut R, Siritaratiwat W, Mato L, Eungpinichpong W, Janyacharoen T. Effect of yoga on the menstrual pain, physical fitness, and quality of life of young women with primary dysmenorrhea. J Bodyw Mov Ther. 2017 Oct;21(4):840-846. doi: 10.1016/j.jbmt.2017.01.014. Epub 2017 Feb 7. PMID 29037637
- [Background] Kirca N, Celik AS. The effect of yoga on pain level in primary dysmenorrhea. Health Care Women Int. 2023 May;44(5):601-620. doi: 10.1080/07399332.2021.1958818. Epub 2021 Sep 17. PMID 34534030
- [Background] Rakhshaee Z. Effect of three yoga poses (cobra, cat and fish poses) in women with primary dysmenorrhea: a randomized clinical trial. J Pediatr Adolesc Gynecol. 2011 Aug;24(4):192-6. doi: 10.1016/j.jpag.2011.01.059. Epub 2011 Apr 21. PMID 21514190
- [Background] Yang NY, Kim SD. Effects of a Yoga Program on Menstrual Cramps and Menstrual Distress in Undergraduate Students with Primary Dysmenorrhea: A Single-Blind, Randomized Controlled Trial. J Altern Complement Med. 2016 Sep;22(9):732-8. doi: 10.1089/acm.2016.0058. Epub 2016 Jun 17. PMID 27315239
- [Background] Gunebakan O, Acar M. The effect of tele-yoga training in healthy women on menstrual symptoms, quality of life, anxiety-depression level, body awareness, and self-esteem during COVID-19 pandemic. Ir J Med Sci. 2023 Feb;192(1):467-479. doi: 10.1007/s11845-022-02985-0. Epub 2022 Mar 24. PMID 35332504
- [Background] Oksuz S, Unal E. The effect of the clinical pilates exercises on kinesiophobia and other symptoms related to osteoporosis: Randomised controlled trial. Complement Ther Clin Pract. 2017 Feb;26:68-72. doi: 10.1016/j.ctcp.2016.12.001. Epub 2016 Dec 8. PMID 28107853